CLINICAL TRIAL: NCT05241509
Title: Biochemical Efficacy of Cymbopogon Citratus Gel as Local Drug Delivery Agent in Reducing Matrix Metalloproteinase-8 Levels Intra-crevicularly in the Treatment of Stage II Periodontitis: A Randomized Controlled Clinical Trial
Brief Title: Cymbopogon Citratus Gel as Local Drug Delivery Agent in Reducing Matrix Metalloproteinase-8 Levels Intra-crevicularly in the Treatment of Stage II Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Souzy Kamal (Other)
Responsible Party: Sponsor-Investigator, Souzy Kamal, lecturer of oral medicine, periodontology, oral diagnosis and radiology, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lemon grass oil
Record Dates: First submitted 2022-01-27; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Periodontitis Chronic Generalized Moderate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group I (test) (Experimental): included twenty patients treated with SRP and intrapocket application of 2% lemongrass oil gel.
  Interventions: Drug: Cymbopogon citratus (lemongrass) oil gel
- Group II (control) (Placebo Comparator): included twenty treated with SRP and intrapocket application of placebo gel.
  Interventions: Drug: Cymbopogon citratus (lemongrass) oil gel

INTERVENTIONS:
Drug: Cymbopogon citratus (lemongrass) oil gel — Biochemical Efficacy of Cymbopogon Citratus Gel as Local Drug Delivery Agent in Reducing Matrix Metalloproteinase-8 Levels Intra-crevicularly in the Treatment of Stage II Periodontitis

SUMMARY:
Background: Phytotherapeutics is widely used nowadays as an adjunct to scaling and root planing (SRP) to modulate inflammatory host response and eradicate microbes. Matrix metalloproteinase-8 (MMP-8) is associated with the onset of inflammation and considered an indicative biomarker to the severity of inflammatory response. Since MMP-8 can be used as a predictive biomarker for treatment response; our research aimed to investigate clinically the effectiveness of intra-pocket application of Cymbopogon citratus (lemongrass oil) gel and biochemically on MMP-8 levels in gingival crevicular fluid (GCF) of stage II periodontitis patients.

Methods: A randomized controlled clinical trial was conducted on forty patients with stage II periodontitis, divided equally into two groups. Group-I (test) was managed by SRP with intra-pocket application of 2% lemongrass oil gel. Group-II (control) was managed by SRP with intra-pocket application of a placebo gel. Periodontal pocket depth (PPD) and clinical attachment loss (CAL) were measured for both groups, before treatment and twelve weeks after. Moreover, GCF was collected from both groups at baseline, one week, and twelve weeks after treatment. Then analysed by Enzyme-linked Assay (ELISA) technique.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy individuals of both sexes having moderate periodontitis (stage II), CAL 3-4mm, with an age ranging from 25 to 45 years old.
* patients with no history of previous periodontal therapy or taken any antibiotic therapy for the past six months

Exclusion Criteria:

* history of smoking, previous adverse reaction to the products (or similar products) used in this study, grade C category that has rapid rate of progression, and pregnant or lactating women

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-06 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2021-12-04 (Actual)

PRIMARY OUTCOMES:
Change in periodontal pocket depth | baseline and after 12 weeks
  the distance between the gingival margin and depth of probing
Change in clinical attachment loss | baseline and after 12 weeks
  the distance between the CEJ and depth of probing
Change in Matrix metalloproteinase-8 level | baseline and after 12 weeks
  Human Matrix metalloproteinase-8 level intracrevicularlly by collection of crevicular fluid sample

CONTACTS AND LOCATIONS:
Overall Officials: Souzy K. Anwar, Ph.D, Principal Investigator — periodontology department. Faculty of dentistry. Alexandria university
Locations (1):
- department of periodontology. Faculty of dentistry. Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF